CLINICAL TRIAL: NCT01963247
Title: Evaluation of the Effectiveness and Clinical Utility of Brain Network Activation (BNA™) Technology in the Management of Sport Related Concussion in Youth Athletes
Brief Title: An Investigator Initiated Study to Evaluate the Effectiveness of Brain Network Activation (BNA™) Technology in the Management of Sport Related Concussion
Status: Completed | Type: Observational
Sponsor: ElMindA Ltd (Industry)
Collaborators: Noran Neurological Clinic (Unknown)
Responsible Party: Sponsor
Other Study IDs: ELM-22
Record Dates: First submitted 2013-10-10; First posted 2013-10-16 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Healthy; Minor Traumatic Brain Injury (TBI)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy Athletes
- Concussed Athletes

SUMMARY:
Currently, there is no direct, reliable, bed-side, and non-invasive method for assessing changes in brain activity associated with concussion. Event Related Potentials (ERPs), which are temporal reflections of the neural mass electrical activity of cells in specific regions of the brain that occur in response to stimuli, may offer such a method, as they provide both a noninvasive and portable measure of brain function. The ERPs provide excellent temporal information, but spatial resolution for ERPs has traditionally been limited. However, by using high-density electroencephalograph (EEG) recording spatial resolution for ERPs is improved significantly. The paradigm for the current study will combine neurophysiological knowledge with mathematical signal processing and pattern recognition methods (BNA™) to temporally and spatially map brain function, connectivity and synchronization.

The proposed study will provide additional evidence for the utility and contribution of the BNA™ test (reflecting temporal and spatial changes in brain activity as well as brain functional connectivity associated with concussion) in concussion management.

The BNA test is basically divided to 3 phases - first EEG data is collected from subjects using an EEG system while the subject is performing a cognitive task in front of a computer. The EEG data is then analyzed using the advanced BNA™ technology. Finally, a report of the BNA™ test is generated.

DETAILED DESCRIPTION:
A single center study evaluating the effectiveness of BNA technology as an objective tool for sport related concussion management in youth athletes' populations.

The study will include 150 athletes from Minnesota Youth Hockey Programs. Subjects enrolled in this study will undergo a screening and baseline pre season visit and follow up visit/s.

1. Follow-up testing for concussed athletes - Concussed athletes will complete a series of post concussion follow up visits. Each will consist of BNA™ test, ImPACT™ test, and exam by neurologist or neurology nurse practitioner. The first visit will be within 72 hours of injury and re-evaluations will occur weekly until BNA has normalized AND subject is asymptomatic. Subject may return to play at that point and subject will have a final additional BNA™ test one week after the athlete returns to full activity. If participant is still symptomatic and/or BNA is still abnormal at 6 weeks reevaluations go to every 2 weeks for up to three months or clearing of symptoms AND normal BNA™. If not back to baseline at three months, monthly reevaluations until study completion.
2. Follow up visit for non-concussed athletes - non-concussed athletes will complete a follow up visit upon completion of the sport season.

ELIGIBILITY:
Inclusion Criteria:

* Male athletes
* aged 11-15
* enrolled in selected Minnesota Youth Hockey Programs

Exclusion Criteria:

* Self-reported history of central nervous system injury or disease (examples will include, but will not be limited to, moderate or severe traumatic brain injury (TBI with a Glasgow Coma Scale < 13), epilepsy, seizures, brain surgery, or any positive neuroimaging results)
* Active head lice infection, open scalp wound
* Deafness, and/or blindness
* A concussion within prior six months
* Residual symptoms or deficits related to a previous concussion
* Long and thick hair that prevents the proper administration of an EEG cap.

Ages: 11 Years to 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 150 male athletes enrolled in Minnesota Youth Hockey Programs, aged 11-15 years.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
changes in BNA™ measures during the sport season | 1 year
  Consistency or changes in BNA™ measures during and after the sport season in both concussed and non concussed athletes compared to pre season BNA™ baseline measures.
Correlation of the BNA measures during the sport season in concussed athletes to the clinical diagnosis, symptom scores and the ImPACT test results. | 1 year
  Correlation of the BNA measures during the sport season in concussed athletes to the clinical diagnosis, symptom scores and the ImPACT test results.

CONTACTS AND LOCATIONS:
Overall Officials: Steven s Lebow, MD, Principal Investigator — Noran Neurological Clinic
Locations (1):
- Noran Neurological Clinic, Minneapolis, Minnesota, United States